CLINICAL TRIAL: NCT01268527
Title: A 12-Day Randomized, Blinded, Vehicle and Active Comparator-Controlled Study to Determine the Efficacy and Safety of Six Concentrations of Topical E6201 Gel in Subjects With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: E6201-E044-204; 2009-014815-11 (EudraCT Number)
Record Dates: First submitted 2010-11-15; First posted 2010-12-31 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis vulgaris
MeSH Terms: interventions — 14-(ethylamino)-8,9,16-trihydroxy-3,4-dimethyl-3,4,9,19-tetrahydro-1H-2-benzoxacyclotetradecine-1,7(8H)-dione; Gels; calcipotriene

ARMS (2):
- Cohort 1 (Experimental): Three concentrations of E6201 topical gel (0.03%, 0.1%, and 0.2%) and active comparator, calcipotriene cream (0.005%), were applied once daily for 12 days to specific test fields determined at Baseline. The 3 concentrations of E6201 gel were dosed first in Cohort 1 to establish the safety and tolerability prior to dosing in Cohort 2.
  Interventions: Drug: 0.03% E6201; Drug: 0.1% E6201; Drug: 0.2% E6201; Other: Placebo - 0.03% gel vehicle; Other: Placebo - 0.1% gel vehicle; Other: Placebo - 0.2% gel vehicle; Drug: Calcipotriene
- Cohort 2 (Experimental): Three concentrations of E6201 topical gel (0.005%, 0.01%, and 0.05%) and active comparator, calcipotriene cream (0.005%), were applied once daily for 12 days to specific test fields determined at Baseline. Cohort 2 participants were not dosed until all participants in Cohort 1 completed treatment and safety data were collected and evaluated.
  Interventions: Drug: 0.005% E6201; Drug: 0.01% E6201; Drug: 0.05% E6201; Other: Placebo - 0.05% gel vehicle; Other: Placebo - 0.01% gel vehicle; Drug: Calcipotriene

INTERVENTIONS:
Drug: 0.03% E6201 — Topical 0.03% E6201 gel was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 1
Drug: 0.1% E6201 — Topical 0.1% E6201 gel was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 1
Drug: 0.2% E6201 — Topical 0.2% E6201 gel was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 1
Drug: 0.005% E6201 — Topical 0.005% E6201 gel was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 2
Drug: 0.01% E6201 — Topical 0.01% E6201 gel was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 2
Drug: 0.05% E6201 — Topical 0.05% E6201 gel was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 2
Other: Placebo - 0.03% gel vehicle — Topical 0.03% gel vehicle (negative control) was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 1
Other: Placebo - 0.1% gel vehicle — Topical 0.1% gel vehicle (negative control) was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 1
Other: Placebo - 0.2% gel vehicle — Topical 0.2% gel vehicle (negative control) was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 1
Other: Placebo - 0.05% gel vehicle — Topical 0.005% gel vehicle (negative control) was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 2
Other: Placebo - 0.01% gel vehicle — Topical 0.01% gel vehicle (negative control) was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 2
Other: Placebo - 0.05% gel vehicle — Topical 0.05% gel vehicle (negative control) was applied once daily to individual specific regions of the psoriatic plaque.
  Arms: Cohort 2
Drug: Calcipotriene — Topical 0.005% calcipotriene (positive control) was applied once daily to individual specific regions of the psoriatic plaque.
  Other Names: Daivonex

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, tolerability and the concentration/response relationship of E6201 in subjects with psoriasis vulgaris.

DETAILED DESCRIPTION:
This is a single center, randomized, blinded, intra-individual comparison in two sequential cohorts of 15 subjects each (30 subjects in total) in an outpatient setting, in which each subject simultaneously receives five topical treatments (3 active, 1 vehicle, and 1 positive control) within one or two psoriatic plaques. Treatments consisted of 3 concentrations of E6201 gel, a negative control (gel vehicle), and a positive control (0.005% calcipotriene cream). The different concentrations of E6201 gel and vehicle control were double-blinded, while the calciprotriene cream was single-blinded. Cohort 2 participants were not dosed until all participants in Cohort 1 completed treatment and safety data were collected and evaluated.

ELIGIBILITY:
Inclusion:

* Chronic stable plaque psoriasis with one or two stable psoriatic plaques(s) suitable in size and location for five separate treatment fields to be assessed within it.
* Males and females aged between 18 and 75 years of age
* The general physical examination should be normal (excluding the skin examination for psoriasis) unless the Investigator considers an abnormality not to be clinically significant with regard to the study
* Females of childbearing potential must have a negative serum beta-human chorionic gonadotropin at Visit 1 (Screening) and a negative urine pregnancy test prior to starting study drug(s) (Visit 2). Female subjects of childbearing potential must agree to be abstinent or to use a highly effective method of contraception throughout the study period and for 30 days after the last dose of study drug.
* Provide written informed consent
* Willing and able to comply with all aspects of the protocol

Exclusion:

* Any clinically significant skin diseases other then chronic stable plaque psoriasis
* Other types of psoriasis than chronic stable plaque variant eg, guttate, pustular, erythodermic, etc
* An unstable course of the disease defined as flare(s) in the previous month
* Subjects who used any concommitant topical treatment for the psoriatic plaque(s) to be studied (other than emollients or salicylic acid) within 8 weeks before the Baseline visit eg corticosteroids or topical immunomodulators, anthralin (dithranil), vitamin D derivatives, ultraviolet-light therapy including sunbathing , or retinoids.
* Subjects who used any of the following systemic treatments within 12 weeks before the Baseline visit eg: corticosteroids or adrenocorticotrophic hormone analogs, retinoids such as acitretin or isotretinoin, cyclosporin, interferon, methotrexate, other immuno-suppressive/immunomodulating drugs, psoralen and ultraviolet A therapy, or biologics
* Subjects planning on significant exposure to sun (sun-bathing)
* Treatment with systemic or locally acting medications which might counter or influence the study aim (eg monoamine oxidase inhibitors, anti-epileptic drugs, anti-psychotic drugs) or medications which are known to provoke or aggravate psoriasis, eg Beta-blockers, antimalarial drugs, and lithium within two weeks before the Baseline visit
* Subject is a dependent person, ie, a relative/family member of the Investigator and/or is a member of the Investigator's staff
* Clinical study participation with any investigational drug less than 30 days prior to study entry or planning to receive an investigational drug during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03-15 (Actual); Primary Completion 2010-12-11 (Actual); Study Completion 2010-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mercer, Study Director — Eisai Limited
Locations (1):
- Bioskin GmbH, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Three concentrations of E6201 topical gel (0.03%, 0.1%, and 0.2%) and active comparator, calcipotriene cream (0.005%), were applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site using separate tuberculin syringes that were filled with approximately 200 uL of each concentration of study treatment and comparator. Prior to each new application, remaining preparation residues were removed by gently cleansing each test field with a separate soft tissue. The fields to be treated were done in an occlusive manner for a treatment period of 12 days. Application time was to be kept as close as possible to the baseline application time, and was not to differ by more than +/- 4 hours. The 3 concentrations of E6201 gel were dosed first in Cohort 1 to establish the safety and tolerability prior to dosing in Cohort 2.
- Cohort 2: Three concentrations of E6201 topical gel (0.005%, 0.01%, and 0.05%) and active comparator, calcipotriene cream (0.005%), were applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described for Cohort 1. Cohort 2 participants were not dosed until all participants in Cohort 1 completed treatment and safety data were collected and evaluated.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one application of at least one study treatment and had at least one postdose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 47.4 (12.44) | 50.6 (7.01) | 49.0 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Summary Statistics and Primary Pairwise Comparison (Vehicle-E6201) of Area Under the Curve (AUC) for the Baseline-Corrected Thickness of the Psoriatic Infiltrate
Description: The AUC was based on the baseline-corrected thickness of the psoriatic infiltrate (20 megahertz (MHz) Sonographic measurement) at specified days for each treatment field calculated by applying the linear trapezoidal rule. Sonographic measurements were performed using a 20 MHz high-frequency sonograph. Serial A-scans were composed and represented on a monitor as a section of the skin. A lateral resolution of approximately 200 um and an axial resolution of 80 um were possible. Dependent on the echo patterns, components of the epidermis, dermis, and subcutis were represented. Therefore, exact measurement of skin thickness was possible. The inflammatory psoriatic infiltrate was seen as a clearly definable echo lucent band below the entrance echo. The thickness of the echo lucent psoriatic band was determined. The thickness was measured in micrometers (um) and was denoted as T.
Time Frame: Day 0 (Baseline), Day 8 (Visit 10), and Day 12 (End of Treatment)
Population: Full analysis population (Intent-to-treat population) included all randomized participants who received at least one application of at least one study treatment and had at least one postbaseline efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: um.day
Groups:
- Daivonex (Calcipotriene Cream): Daivonex (calcipotriene cream) at 0.005% was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site using a tuberculin syringe that was filled with approximately 200 uL of Daivonex. Prior to each new application, remaining preparation residues were removed by gently cleansing each test field with a separate soft tissue. The fields to be treated were done in an occlusive manner for a treatment period of 12 days. Application time was to be kept as close as possible to the baseline application time, and was not to differ by more than +/- 4 hours.
- E6201 Vehicle: E6201 vehicle was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
- 0.005% E6201 Gel: E6201 gel (0.005%) was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
- 0.01% E6201 Gel: E6201 gel (0.01%) was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
- 0.03% E6201 Gel: E6201 gel (0.03%) was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
- 0.05% E6201 Gel: E6201 gel (0.05%) was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
- 0.1% E6201 Gel: E6201 gel (0.1%) was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
- 0.2% E6201 Gel: E6201 gel (0.2%) was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
Arm/Group | Daivonex (Calcipotriene Cream) | E6201 Vehicle | 0.005% E6201 Gel | 0.01% E6201 Gel | 0.03% E6201 Gel | 0.05% E6201 Gel | 0.1% E6201 Gel | 0.2% E6201 Gel
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 15 | 15 | 6 | 6
um.day | -1449.2 [-1660.0 to -1238.4] | 17.0 [-64.3 to 98.3] | -694.4 [-1108.0 to -280.8] | -1102.8 [-1351.8 to -853.8] | -763.1 [-1548.2 to 22.1] | -1758.2 [-2134.3 to -1382.1] | -904.4 [-1303.4 to -505.4] | -920.8 [-1588.3 to -253.3]
Statistical Analysis 1: Comparison: E6201 Vehicle vs 0.005% E6201 Gel; The following hypotheses were based on the Full Analysis Population: null Hypothesis and alternative hypothesis. P values, Least Squares Means (LSM), and Confidence Intervals (CI) were obtained from ANCOVA model with factors for treatment and baseline psoriatic infiltrate thickness as a continuous covariate; Test type: Superiority; p = 0.0038, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 711.4, 95% CI 2-sided [292.5 to 1130.3]
Statistical Analysis 2: Comparison: E6201 Vehicle vs 0.01% E6201 Gel; The following hypotheses were based on the Full Analysis Population: null Hypothesis and alternative hypothesis. P values, LSM, and CI were obtained from ANCOVA model with factors for treatment and baseline psoriatic infiltrate thickness as a continuous covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 1119.8, 95% CI 2-sided [858.9 to 1380.6]
Statistical Analysis 3: Comparison: E6201 Vehicle vs 0.03% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0523, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 780.0, 95% CI 2-sided [-8.5 to 1568.5]
Statistical Analysis 4: Comparison: E6201 Vehicle vs 0.05% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 1775.1, 95% CI 2-sided [1392.3 to 2158.0]
Statistical Analysis 5: Comparison: E6201 Vehicle vs 0.1% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0002, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 921.4, 95% CI 2-sided [515.7 to 1327.1]
Statistical Analysis 6: Comparison: E6201 Vehicle vs 0.2% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0115, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 937.8, 95% CI 2-sided [267.6 to 1607.9]

2. Secondary Outcome: Change in Thickness of the Psoriatic Infiltrate From Baseline to End of Treatment (Day 12/Discontinuation)
Description: Psoriatic infiltrate thickness was determined by 20 MHz Sonographic measurements using a 20 MHz high-frequency sonograph. Serial-A scans were composed and represented on a monitor as a section of the skin. A lateral resolution of approximately 200 um and an axial resolution of 80 um were possible. Dependent on the echo patterns, components of the epidermis, dermis, and subcutis were represented. Therefore exact measurement of the skin thickness was possible. The inflammatory psoriatic infiltrate was seen as a clearly definable echo lucent back below the entrance echo. The thickness of the echo lucent psoriatic band was determined. Comparisons were made with the untreated plaque(s) beneath the hydrocolloid dressing. Baseline was defined as Visit 2 (Day 0). Least Squares Means (LSM) and Confidence Intervals (CI) were obtained from ANCOVA model with factors for treatment and baseline psoriatic infiltrate thickness as a continuous covariate.
Time Frame: Day 12/Discontinuation (Visit 14/End of Treatment)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: um
Groups:
- E6201 Vehicle: E6201-vehicle was applied once daily for 12 days to specific test fields determined at Baseline. Study treatments were applied at the research unit by designated personnel of the investigational site in the same manner as described earlier.
Arm/Group | Daivonex (Calcipotriene Cream) | E6201 Vehicle | 0.005% E6201 Gel | 0.01% E6201 Gel | 0.03% E6201 Gel | 0.05% E6201 Gel | 0.1% E6201 Gel | 0.2% E6201 Gel
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 15 | 15 | 6 | 6
um | -205.3 [-239.2 to -171.4] | 7.1 [-32.2 to 46.3] | -94.4 [-154.5 to -34.3] | -175.3 [-206.5 to -144.1] | -162.4 [-194.1 to -130.7] | -239.5 [-295.8 to -183.2] | -125.2 [-202.3 to -48.2] | -137.9 [-218.3 to -57.6]
Statistical Analysis 1: Comparison: E6201 Vehicle vs 0.005% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0042, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 101.5, 95% CI 2-sided [36.0 to 167.0]
Statistical Analysis 2: Comparison: E6201 Vehicle vs 0.01% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 182.4, 95% CI 2-sided [140.3 to 224.4]
Statistical Analysis 3: Comparison: E6201 Vehicle vs 0.03% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 169.5, 95% CI 2-sided [127.4 to 211.5]
Statistical Analysis 4: Comparison: E6201 Vehicle vs 0.05% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 246.6, 95% CI 2-sided [185.0 to 308.1]
Statistical Analysis 5: Comparison: E6201 Vehicle vs 0.1% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0043, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 132.3, 95% CI 2-sided [53.9 to 210.7]
Statistical Analysis 6: Comparison: E6201 Vehicle vs 0.2% E6201 Gel; The following hypotheses were based on the Full Analysis Population: null Hypothesis and alternative hypothesis. P values, LSM) and CI were obtained from ANCOVA model with factors for treatment and baseline psoriatic infiltrate thickness as a continuous covariate; Test type: Superiority; p = 0.0036, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 145.0, 95% CI 2-sided [64.2 to 225.8]

3. Secondary Outcome: Change in Thickness of the Psoriatic Infiltrate From Baseline to Day 8
Description: Psoriatic infiltrate thickness was determined by 20 MHz Sonographic measurements using a 20 MHz high-frequency sonograph. Serial-A scans were composed and represented on a monitor as a section of the skin. A lateral resolution of approximately 200 um and an axial resolution of 80 um were possible. Dependent on the echo patterns, components of the epidermis, dermis, and subcutis were represented. Therefore exact measurement of the skin thickness was possible. The inflammatory psoriatic infiltrate was seen as a clearly definable echo lucent back below the entrance echo. The thickness of the echo lucent psoriatic band was determined. Comparisons were made with the untreated plaque(s) beneath the hydrocolloid dressing. Baseline was defined as Visit 2 (Day 0). LSM and CI were obtained from ANCOVA model with factors for treatment and baseline psoriatic infiltrate thickness as a continuous covariate.
Time Frame: Day 8 (Visit 10)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: um
Arm/Group | Daivonex (Calcipotriene Cream) | E6201 Vehicle | 0.005% E6201 Gel | 0.01% E6201 Gel | 0.03% E6201 Gel | 0.05% E6201 Gel | 0.1% E6201 Gel | 0.2% E6201 Gel
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 15 | 15 | 6 | 6
um | -151.7 [-215.1 to -88.3] | 17.3 [-20.2 to 54.8] | -63.4 [-110.3 to -16.5] | -110.7 [-147.3 to -74.0] | -92.9 [-200.1 to 14.3] | -190.3 [-243.6 to -136.9] | -108.0 [-162.9 to -53.1] | -102.7 [-172.6 to -32.9]
Statistical Analysis 1: Comparison: E6201 Vehicle vs 0.005% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0013, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 80.7, 95% CI 2-sided [34.6 to 126.7]
Statistical Analysis 2: Comparison: E6201 Vehicle vs 0.01% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 127.9, 95% CI 2-sided [92.4 to 163.5]
Statistical Analysis 3: Comparison: E6201 Vehicle vs 0.03% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0458, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 110.2, 95% CI 2-sided [2.4 to 218.0]
Statistical Analysis 4: Comparison: E6201 Vehicle vs 0.05% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 207.5, 95% CI 2-sided [155.2 to 259.9]
Statistical Analysis 5: Comparison: E6201 Vehicle vs 0.1% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0003, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 125.3, 95% CI 2-sided [71.5 to 179.0]
Statistical Analysis 6: Comparison: E6201 Vehicle vs 0.2% E6201 Gel; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0029, ANCOVA; Difference in LSM (vehicle - E6201 gel) = 128.6, 95% CI 2-sided [93.9 to 163.3]

4. Secondary Outcome: Clinical (Global) Assessment of Efficacy at Day 12/Discontinuation
Description: Clinical (global) assessment of the test fields was performed using a 5-point score: -1 = worsened, 0 = unchanged (no effect), 1 = slight improvement, 2 = clear improvement but not completely healed, and 3 = completely healed. Comparisons were made with the untreated plaque(s) beneath the hydrocolloid dressing. Clinically apparent differences in erythema and infiltration contributed to the global assessment. Baseline was defined as Visit 2 (Day 0).
Time Frame: Day 12/Discontinuation (Visit 14/End of Treatment)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Daivonex (Calcipotriene Cream) | E6201 Vehicle | 0.005% E6201 Gel | 0.01% E6201 Gel | 0.03% E6201 Gel | 0.05% E6201 Gel | 0.1% E6201 Gel | 0.2% E6201 Gel
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 15 | 15 | 6 | 6
Percentage of participants
  Worsened | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unchanged (no effect) | 6.7 | 90.0 | 20.0 | 0 | 6.7 | 0 | 0 | 0
  Slight improvement | 56.7 | 10.0 | 66.7 | 33.3 | 46.7 | 13.3 | 83.3 | 83.3
  Clear improvement but not completely healed | 33.3 | 0 | 13.3 | 66.7 | 46.7 | 86.7 | 16.7 | 0
  Completely healed | 3.3 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7

5. Secondary Outcome: Clinical (Global) Assessment of Efficacy on Day 8
Description: as for outcome 4
Time Frame: Day 8 (Visit 10)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Daivonex (Calcipotriene Cream) | E6201 Vehicle | 0.005% E6201 Gel | 0.01% E6201 Gel | 0.03% E6201 Gel | 0.05% E6201 Gel | 0.1% E6201 Gel | 0.2% E6201 Gel
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 15 | 15 | 6 | 6
Percentage of participants
  Worsened | 3.3 | 3.3 | 0 | 0 | 6.7 | 0 | 0 | 0
  Unchanged (no effect) | 20.0 | 90.0 | 33.3 | 6.7 | 6.7 | 0 | 16.7 | 0
  Slight improvement | 46.7 | 6.7 | 66.7 | 53.3 | 60.0 | 13.3 | 83.3 | 100
  Clear improvement but not completely healed | 30.0 | 0 | 0 | 40.0 | 26.7 | 86.7 | 0 | 0
  Completely healed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Overview of Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as an adverse event (AE) that emerged during treatment, having been absent at pretreatment (baseline), or re-emerged during treatment, having been present at baseline but stopped prior to treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. Safety variables included TEAEs including skin reactions, diascopy and biopsy findings, clinical laboratory parameters, vital signs, and physical examinations. For Cohort 2, special attention was given to a close, daily monitoring of the application site for signs of skin irritation. Any suspected ecchymoses or petechiae were to be followed up with a diascopy test that was to be documented with digital photographs. Any positive diascopy test was to be followed up by biopsy for skin ultrastructural analysis (if agreed to by the participant, sponsor, and investigator). Few adverse events occurred in more than one treatment group.
Time Frame: From first dose of study treatment up to 30 days after the last dose, or until resolution, whichever came first, or up to approximately 10 months.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Daivonex (Calcipotriene Cream) | E6201 Vehicle | 0.005% E6201 Gel | 0.01% E6201 Gel | 0.03% E6201 Gel | 0.05% E6201 Gel | 0.1% E6201 Gel | 0.2% E6201 Gel
Number analyzed (Participants) | 30 | 30 | 15 | 15 | 15 | 15 | 6 | 6
Percentage of participants
  TEAEs | 3 | 1 | 0 | 0 | 4 | 5 | 6 | 6
  Treatment-related TEAEs | 3 | 1 | 0 | 0 | 4 | 5 | 6 | 6
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to study treatment withdrawal | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  TEAEs leading to study treatment dose decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to study treatment interruption | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 30 days after the last dose, or until resolution, whichever came first, or up to approximately 10 months.
Description: Treatment-emergent adverse events (TEAEs) were collected and defined as an AE that emerged during treatment, having been absent at pretreatment, or re-emerged during treatment, having been present at baseline but stopped prior to treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. Few adverse events occurred in more than one treatment group.
Arm/Group | Daivonex (Calcipotriene Cream) | E6201 Vehicle | 0.005% E6201 Gel | 0.01% E6201 Gel | 0.03% E6201 Gel | 0.05% E6201 Gel | 0.1% E6201 Gel | 0.2% E6201 Gel
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/15 | 0/15 | 0/15 | 0/15 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/15 | 0/15 | 0/15 | 0/15 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/30 | 1/30 | 0/15 | 0/15 | 4/15 | 5/15 | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daivonex (Calcipotriene Cream) (N=30) | E6201 Vehicle (N=30) | 0.005% E6201 Gel (N=15) | 0.01% E6201 Gel (N=15) | 0.03% E6201 Gel (N=15) | 0.05% E6201 Gel (N=15) | 0.1% E6201 Gel (N=6) | 0.2% E6201 Gel (N=6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 5 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5
Lividity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other